CLINICAL TRIAL: NCT03752788
Title: Dual-Task Training With Variable Priority Instructional Sets Improve the Gait Parameters in Patients With Chronic Stroke
Brief Title: Dual-Task Training With Different Priority Instructional Sets on the Gait Parameters in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRC-2017-005
Record Dates: First submitted 2018-11-19; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Stroke; Middle Cerebral Artery Stroke; Chronic Stroke
Keywords: Stroke; Gait velocity; Stride length; Step length; Balance training; Dual task; Institutional priority sets
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task Training Fixed Priority (Experimental): Dual-task Training with fixed priority instructional set for four weeks. Balance training sessions of 45 minutes per day, 3 times a week for four weeks, so as to complete 9-12 hours of training warm-up improve the balance performance. This included 12 repetitions in each session for 30 minutes after a 10-minutes warm up.
  Attention was focused on both postural and cognitive tasks throughout this session. In postural tasks, subjects were instructed to perform the following: walk narrow base of support with a cognitive task of counting backward by three walk narrow base of support with cognitive task of count forward by three, walk narrow base of support, step, sideways, backward avoiding the obstacles (holding a basket) with cognitive task to remember words.
  Interventions: Behavioral: Dual-task Training Fixed Priority
- Dual-task Training Variable Priority (Active Comparator): Dual-task Training with variable priority instructional set for four weeks. Balance training sessions of 45 minutes per day, 3 times a week for four weeks, so as to complete 9-12 hours of training warm-up improve the balance performance. This included 12 repetitions in each session for 30 minutes after a 10-minutes warm up.
  During the first half of the training session, attention was focused on postural tasks, while during the remaining half of the session, attention was focused on cognitive tasks.
  Interventions: Behavioral: Dual-task Training Variable Priority

INTERVENTIONS:
Behavioral: Dual-task Training Fixed Priority — Dual-task training fixed priority instructional set for four weeks. Balance training sessions of 45 minutes per day, 3 times a week for four weeks, so as to complete 9-12 hours of training warm-up improve the balance performance. This included 12 repetitions in each session for 30 minutes after a 10-minutes warm up.
  Attention was focused on both postural and cognitive tasks throughout this session. In postural tasks, subjects were instructed to perform the following: walk narrow base of support with a cognitive task of counting backward by three walk narrow base of support with cognitive task of count forward by three, walk narrow base of support, step, sideways, backward avoiding the obstacles (holding a basket) with cognitive task to remember words.
  Arms: Dual-task Training Fixed Priority
Behavioral: Dual-task Training Variable Priority — Dual-task training variable priority instructional set for four weeks. Balance training sessions of 45 minutes per day, 3 times a week for four weeks, so as to complete 9-12 hours of training warm-up improve the balance performance. This included 12 repetitions in each session for 30 minutes after a 10-minutes warm up.
  During the first half of the training session, attention was focused on postural tasks, while during the remaining half of the session, attention was focused on cognitive tasks.
  Arms: Dual-task Training Variable Priority

SUMMARY:
Balance is controlled through a complex process involving sensory, visual, vestibular and cerebral functioning which get affected by various neurological disorders such as in stroke. Different types of exercises are designed to target to cope up with the imbalance developed due to these neurological disorders. This study aimed to compare the efficacy of dual-task training using two different priority instructional sets in improving gait parameters such as self-selected velocity, fast speed, step length, and stride length in chronic stroke patients.

DETAILED DESCRIPTION:
Balance is controlled through a complex process involving sensory, visual, vestibular and cerebral functioning which get affected by various neurological disorders such as in stroke. Different types of exercises are designed to target to cope up with the imbalance developed due to these neurological disorders. This study aimed to compare the efficacy of dual-task training using two different priority instructional sets in improving gait parameters such as self-selected velocity, fast speed, step length, and stride length in middle cerebral artery chronic stroke patients. A total of thirty middle cerebral artery chronic stroke patients were recruited on the basis of inclusion and exclusion criteria and equally allocated into two groups. Group 1 received dual-task training with fixed priority instructional sets for four weeks and group 2 received dual-task training with variable priority instructional sets for four weeks. The outcome was assessed using a 10-meter walk test and the comparison of footprints on the walkway paper before and after training.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosed case of middle cerebral artery chronic stroke made by a neurologist and verified using CT/MRI
* Exhibited the age between 45 and 65 years
* Ability to walk 10 meters without assistance
* Their stroke onset within 12 months prior to the study and
* Scored greater than 24 on Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* Participants had neurological conditions other than stroke
* Uncontrolled hearing or visual and vestibular impairment
* Took more than 15 seconds on Timed Up & Go (TUG) test
* Had lower extremity amputation
* A case of diagnosed speech-language impairment (not able to respond verbally to auditory stimuli) by a speech-language pathologist and noticed their concurrent participation in another clinical trial

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
10-meter walk test | Change from Baseline 10-meter Walk Test scores at 4-Weeks
  It is used to evaluate gate parameters such as gait velocity (self-selected velocity and fast velocity, step length and stride length ) in patients with chronic stroke.

SECONDARY OUTCOMES:
Mini-mental state examination (MMSE) or Folstein test | Before the study intervention
  It is used to to determine any impaired cognition that would affect the ability of the participant with stroke to follow instructions.
Timed Up & Go (TUG) test | Before the study intervention
  It is used to identify the patient's mobility with respect to healthy elderly subjects, such as the gait parameters and walking endurance in subjects with chronic stroke.The TUG score correlates with gait speed, balance, functional level, ability to go out, and this score can change over time.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Principal Investigator — Rehabilitation Research Chair
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
Undecided